CLINICAL TRIAL: NCT06806774
Title: Reliability and Validity of the Glittre Activities of Daily Living Test in Children and Adolescents With Juvenile Idiopathic Arthritis
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sinan Buran, Research Assistant, Hacettepe University
Other Study IDs: SBA 24/999
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Juvenile Idiopathic Arthritis (JIA)
Keywords: activities of daily living; reliability; validity; juvenile idiopathic arthritis; functional capacity
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Juvenile Idiopathic Arthritis (JIA)

SUMMARY:
Juvenile Idiopathic Arthritis (JIA) is children's most common inflammatory rheumatic disease. The International League of Associations for Rheumatology (ILAR) defines it as a chronic arthritis condition that begins before the age of 16 lasts for six weeks or more, and has an unknown cause. Despite the gains made in the management of the disease of individuals with JIA with modern medical treatment methods, the physical and psychosocial problems caused by chronic inflammation negatively affect the daily living activities of individuals with JIA. On the other hand, in the JIA Core Set created by Outcome Measures in Rheumatology (OMERACT) in 2018, activities of daily living were included as a "mandatory area that should be evaluated in all studies." Therefore, to ensure that individuals with JIA reach a state of complete well-being, multi-interdisciplinary health professionals are expected to address the activities of daily living, identify the factors that limit these activities, and create intervention plans for the factors to be determined. The literature shows that the daily living activities of patients with JIA are addressed with a limited number of subjective measurement tools. However, these methods have disadvantages due to their subjectivity. In this case, objective measurement methods are needed to quantify the physical performance of patients with JIA in terms of their daily living activities. The Glittre Activities of Daily Living Test, initially developed by selecting activities similar to daily living activities to evaluate functional capacity in pulmonary diseases, has the potential to address this gap. Since the activities in the test require using both the lower and upper extremities, it has the advantage of reflecting functional capacity and providing information about performance in daily life activities. Although it has potential, the Glittre Activities of Daily Living Test needs appropriate psychometric properties for clinical settings and research for JIA patients. To our knowledge, no studies have been conducted in the current literature on the validity and reliability of the Glittre Activities of Daily Living Test in JIA patients. Therefore, this study aimed to evaluate the test-retest reliability, construct validity, and minimum detectable change of the Glittre Activities of Daily Living Test in assessing activities of daily living in children and adolescents with JIA.

DETAILED DESCRIPTION:
Juvenile Idiopathic Arthritis (JIA) is children's most common inflammatory rheumatic disease. The International League of Associations for Rheumatology (ILAR) defines it as a chronic arthritis condition that begins before age 16, lasts six weeks or more, and has an unknown cause. Despite the gains made in the management of JIA patients with modern medical treatment methods, there are physical and psychosocial problems caused by chronic inflammation. While chronic pain, disease activity, fatigue, and musculoskeletal problems constitute the physical dimension of these effects, issues such as anxiety, depression, central sensitization of pain, decreased peer interaction, physical activity, and school participation constitute the psychosocial dimension. In a study that addressed these biopsychosocial problems holistically within the framework of the International Classification of Functioning Disability and Health - Children and Youth (ICF-CY), it was emphasized that the daily living activities of individuals diagnosed with JIA were negatively affected, resulting in participation restrictions in various environments. On the other hand, in the JIA Core Set created by Outcome Measures in Rheumatology (OMERACT) in 2018, activities of daily living were included as a "mandatory area that should be evaluated in all studies." Therefore, to ensure that patients with JIA reach a state of complete well-being, multidisciplinary health professionals are expected to address the activities of daily living, identify the factors that limit these activities, and create intervention plans for the factors to be determined. The literature shows that the daily living activities of patients with JIA are addressed with a limited number of subjective measurement tools, especially the Childhood Health Assessment Questionnaire (CHAQ). CHAQ, widely used in evaluating daily living activities in pediatric rheumatology, stands out with its advantages, such as being practical, short, easy to score, and providing a commonly spoken language due to its adaptation to many languages. However, CHAQ also has some disadvantages. These disadvantages are that CHAQ is known for its ceiling effect, its subjective aspect, and its relative insensitivity to short-term changes. Physical function is a complex and multidimensional phenomenon associated with the ability to move and perform daily activities. Measuring physical function is essential to provide targets for clinical intervention to reduce impairments and increase participation in activities. By assessing physical function, baseline function can be objectively determined before treatment, which is essential for evaluating the effectiveness of the intervention. Physical function is usually measured with physical performance tests and self-report questionnaires. Physical performance tests quantify performance, as opposed to the perception of performance obtained through self-report questionnaires, thus providing a more objective measure of actual functional capacity. Performance-based measures have theoretical advantages over self-report measures, such as better repeatability, greater sensitivity to change, and less influence by external influences such as culture, language, and education. The "Glittre Activities of Daily Living Test," a physical function-based test that objectively evaluates daily living activities, was initially developed by selecting activities similar to daily living activities to assess functional capacity in Chronic Obstructive Pulmonary Disease. Since the activities in the Glittre Activities of Daily Living Test require using both the lower and upper extremities, the test has the advantages of reflecting functional capacity and providing information about performance in daily living activities. Due to these advantages, reliability and validity studies have been conducted on diseases other than chronic obstructive pulmonary disease, which was the starting point. The Glittre Activities of Daily Living Test rules were initially developed for adult patients and modified because they were unsuitable for the pediatric group. The modified test, the Pediatric Glittre Activities of Daily Living Test, was valid and reliable in children aged 6-14. One of the primary treatment goals is to ensure that patients with JIA maintain their daily living activities. Activities of daily living are also considered an important outcome measure for evaluating the course of the disease and the effectiveness of treatment. When the literature is examined, self-reporting questionnaires are used more frequently to assess the daily living activities of JIA patients, and performance-based standardized measurement methods are used less frequently. When considering the needs of individuals with JIA, the Glittre Activities of Daily Living Test has significant potential in this disease group. However, its psychometric properties must be appropriate in clinical settings and research. To our knowledge, no studies on the validity and reliability of the Glittre Activities of Daily Living Test in JIA patients have been conducted in the current literature. Therefore, this study aimed to evaluate the test-retest reliability, construct validity, and minimum detectable change of the Glittre Test of Activities of Daily Living in assessing activities of daily living in children and adolescents with JIA. Since the test is modified for 6-to 14-year-olds, the "Pediatric Glittre Activities of Daily Living Test" reliability and validity will be assessed in individuals with JIA within this age group. The standard version will be used for JIA patients between 15 and 18.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Juvenile Idiopathic Arthritis (JIA) according to The International League of Associations for Rheumatology (ILAR) classification
* Being between the ages of 8-18
* Volunteering to participate in research

Exclusion Criteria:

* Advanced heart/lung/liver/kidney disease, neurological disease and malignancies
* Having undergone major orthopedic surgery
* Not volunteering to participate in the study

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of individuals with JIA who meet the inclusion criteria at the Department of Pediatrics, Division of Rheumatology, Hacettepe University Faculty of Medicine.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The Glittre Activities of Daily Living Test | Baseline (First Assessment)
  The Glittre Activities of Daily Living Test is widely used in the literature to evaluate activities of daily living based on performance. The test consists of a cycle of standardized activities such as walking, weight-bearing, climbing stairs, and moving objects on shelves. It is a test that takes place over a total distance of 10 m divided into two parts by a ladder. The person completes the test cycle in 5 laps at this distance range. The time it takes for individuals to complete the test and their pre-and post-test heart rate, blood pressure, respiratory frequency, SpO2, and modified Borg Scale, as well as their dyspnea and fatigue levels during exertion, are evaluated. In our study, the Pediatric Glittre Activities of Daily Living Test will be used for individuals diagnosed with JIA between the ages of 8 and 14, and the standard version of the test will be used for JIA patients between the ages of 15 and 18.

SECONDARY OUTCOMES:
Functional Reach Test | Baseline (First assessment)
  The Functional Reach Test is a test that evaluates dynamic balance. The person is asked to stand with their arm at 90̊ flexion and close to the wall without touching it; then, they are instructed to reach forward as far as they can without taking a step. The difference between the start and finish is measured with a tape measure and recorded in centimeters. Three trials are performed; the average is the Functional Reach Test score.
Six Minute Walk Test (6MWT) | Baseline (First Assessment)
  For the 6MWT, individuals are asked to walk in a 30-meter corridor at the maximal speed they can walk without running. During the test, individuals are encouraged with standard expressions. At the end of the test, the distance covered will be recorded in meters. The individuals' pre-test and post-test heart rate, blood pressure, respiratory frequency, SpO2, and modified Borg Scale, as well as dyspnea and fatigue levels during exertion, will be evaluated.
Childhood Health Assessment Questionnaire (CHAQ) | Baseline (First Assessment)
  The CHAQ assesses the functional abilities of children with JIA in activities of daily living. It comprises eight sections (dressing and grooming, arising, eating, walking, hygiene, reaching, griping, and activities) and evaluates pain (0: no pain and 10: extreme pain) and general well-being (0: no problem and 10: extreme problem) using a Visual Analog Scale. The total CHAQ score ranges from 0 to 3 (higher scores reflect low functionality).
Juvenile Arthritis Biopsychosocial Questionnaire (JAB-Q) | Baseline (First Assessment)
  JAB-Q evaluates the problems experienced by both the child and the parent from a biopsychosocial perspective. The scale was developed initially in Turkish. It includes two separate forms for the child (patient) and parent (family) to complete. The child form consists of questions evaluating parameters such as pain intensity, disease activity, joint status, functional assessment, psychosocial status assessment, school status and fatigue, and is scored between 0 and 52 points. The family form includes parameters such as the parent's perception of health and psychosocial status and scores between 0 and 38. Forms can give both total scores and separate scores for subparameters. Higher scores indicate worse results.
Juvenile Arthritis Quality of Life Questionnaire (JAQQ) | Baseline (First Assessment)
  JAQQ, a scale developed for patients with Juvenile Idiopathic Arthritis, consists of 74 items that assess various health domains, including physical functioning, emotional well-being, and general symptoms. The items are categorized into four dimensions related to the child's quality of life: gross motor function, fine motor function, psychosocial function, and systemic symptoms. The questionnaire provides separate scores for these four dimensions and a total score. All scores are scored between 0 and 7. Higher scores indicate a lower quality of life. Doğan et al. conducted the Turkish validity and reliability study of the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sinan Buran, MSc, Principal Investigator — Hacettepe University Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No